CLINICAL TRIAL: NCT05375240
Title: A Randomized, Blank-controlled, Open Label Study of the Safety and Efficacy of Propranolol in Reducing Stroke Associated Pneumonia and Urinary Tract Infection
Brief Title: Propranolol on Post Stroke Immune Status and Infection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Fu-Dong Shi, Professor of Immunology, Neurologist-in-Chief, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2022-YX-001
Record Dates: First submitted 2022-04-19; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Stroke; Cerebrovascular Disorders; Ischemic Stroke; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Cardiovascular Diseases; Propranolol; Beta Blocker; Molecular Mechanisms of Pharmacological Action; Immunologic Factors; Physiological Effects of Drugs
Keywords: Stroke; Propranolol; Infection; Treatment
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Ischemic Stroke; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Cardiovascular Diseases; Infections | interventions — Propranolol; Ceftriaxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blank-control group (No Intervention): Patients will receive standard treatment.
- Oropranolol group (Experimental): Propranolol will be administered at a dose of 10mg*3/day over a course of 7 consecutive days after stroke onset.
  Interventions: Drug: Propranolol
- Propranolol + ceftriaxone group (Experimental): Propranolol will be administered at a dose of 10mg*3/day combined with 2g/day ceftriaxone over a course of 7 consecutive days after stroke onset.
  Interventions: Drug: Propranolol; Drug: Ceftriaxone

INTERVENTIONS:
Drug: Propranolol — Propranolol will be given at a dose of 10 mg orally, 3 times per day, for 7 consecutive days after stroke onset.
  Arms: Oropranolol group; Propranolol + ceftriaxone group
Drug: Ceftriaxone — Intravenously 2.0g/day for 7 consecutive days.
  Arms: Propranolol + ceftriaxone group

SUMMARY:
Stroke-associated pneumonia (SAP) is one of the important risk factors influencing poor outcomes and death in stroke patients. Over the past two decades, accumulating evidence suggests that post-stroke brain injury mobilizes the adrenergic system, which induces post-stroke immunosuppression and SAP. This study is designed to test the safety and efficacy of an adrenergic β-receptor blocker, propranolol, with or without combination of antibiotics, in reducing SAP in stroke patients. The underlying immune mechanisms will be investigated.

DETAILED DESCRIPTION:
Stroke patients meeting the inclusion criteria will be randomly assigned at a 1:1:1 ratio into groups of standard treatment (blank-controlled), propranolol, or propranolol + ceftriaxone.

Patients will be given 10.0mg*3/day oral/nil propranolol alone or combined with 2.0g/day intravenous ceftriaxone over the course of 7 consecutive days. Neurological functions of these patients will be assessed at the baseline, day 7, 14, 30, and 90 after randomization. Head magnetic resonance imaging (MRI) will be performed at baseline and 7 days after randomization. Chest computed tomography (CT) will be performed within 7 days following randomization. Abdomen CT will be performed simultaneously with CT chest to evaluate spleen volume. For patients requiring acute endotracheal intubation upon admission, bronchoalveolar lavage fluid will be harvested at baseline and 7 days post-randomization. For all patients, 15 mL intravenous blood will be collected at baseline, days 3 and 7 after randomization. Bronchoalveolar lavage fluid and blood will be used to explore the peripheral and pulmonary immune status of patients. Urinary tract infection will be evaluated within 14 days based on routine urine test and bacterial culture.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 60 years older and less than 90 years.
2. Onset of new neurological deficits within 24 hours at the time of randomization and propranolol treatment can be initiated within 24 hours of symptom onset.
3. Clinical signs consistent with the diagnosis of stroke, including impairment of language, motor function, cognition, and/or gaze, vision, or neglect.
4. Initial NIHSS score of 11 or greater or Total GCS score (aggregate of verbal, eye, and motor response scores) of 5 or greater and no more than 12 at time of enrollment.
5. MRI or CT scan confirmed stroke.
6. Inability to tolerate normal diet or fluids because of: a. impaired consciousness levels; b. failed clinical bedside swallowing assessment performed by a trained and qualified assessor; c. "nil orally" orders, nasogastric tubes, modified diet or requiring compensatory feeding techniques.
7. TOAST: Large-artery atherosclerosis.
8. Signed and dated informed consent by the subject, legally authorized representative, or surrogate obtained.

Exclusion Criteria:

1. Time of symptom onset that cannot be reliably assessed.
2. Subjects considered as candidates for immediate surgical intervention by the neurosurgery service.
3. Pregnancy or parturition within previous 30 days or active lactation.
4. Coagulation disorders (platelet count less than 50x109/L, elevated baseline APTT or INR>1.3) or use of anti-coagulant drugs within the last 24 hours.
5. Use of beta blockers (propranolol, metoprolol, sotalol, carvedilol, bisoprolol, atenolol, esmolol) or antibiotics within 30 days.
6. Use of reserpine within the last 30 days.
7. Pre-stroke dementia or disability.
8. Admission with any of following signs: 1). Fever>38℃; 2). Signs of pneumonia in chest CT scan; 3). White blood cell count>12000 or <4000 /μL; 4). Cough, sputum or dyspnea; 5). Respiratory rate>25.
9. Severe liver, kidney disease, or malignancy, life expectancy is less than 14 days.
10. Bronchial asthma or COPD.
11. Cardiogenic shock.
12. Severe or acute heart failure.
13. Degree II-III atrioventricular block.
14. Sinus bradycardia (heart rate ≤75/min).
15. Known anergic to propranolol or amoxicillin.
16. Current participation in other interventional clinical trials.
17. Immunosuppressant therapy or known immunosuppression.
18. Inability to undergo neuroimaging with magnetic resonance.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of pneumonia | Up to 7 days
  Stroke-associated pneumonia diagnosed in accordance to a defined algorithm.

SECONDARY OUTCOMES:
Assessment of clinical outcome by National Institute of Healthy Stroke Scale | Up to 90 days
  National Institute of Healthy Stroke Scale(0-42 score),higher scores mean a worse outcome.
Assessment of clinical outcome by modified Barthel Index | Up to 90 days
  Modified Barthel Index（0-100 score),higher scores mean a better outcome.
Assessment of clinical outcome by modified Rankin Scale | Up to 90 days
  Modified Rankin Scale(0-5 score),higher scores mean a worse outcome.
Assessment of clinical outcome by Glasgow Coma Scale | Up to 90 days
  Glasgow Coma Scale(0-15),higher scores mean a better outcome.
Incidence of urinary tract infection | Up to 14 days
  Urinary tract infection diagnosed with defined criteria.
Incidence of sepsis | Up to 14 days
  Sepsis diagnosed with defined criteria.
Alterations of spleen volume | Up to 7 days
  Spleen volume will be evaluated within 7 days via abdomen CT scan.
Single cell sequencing results of immune cells from blood and bronchoalveolar lavage fluid | Up to 7 days
  Single cell sequencing of immune cells from blood and bronchoalveolar lavage fluid will be conducted at baseline and 7 days after stroke onset.
Concentration of soluble protein in blood and bronchoalveolar lavage fluid | Up to 7 days
  Soluble proteins in blood and bronchoalveolar lavage fluid will be evaluated by O-link at baseline and 7 days after stroke onset
Counts of lymphocytes in blood | Up to 7 days
  Counts of lymphocytes will be evaluated by flow cytometry at baseline, day 3, and day 7 post stroke onset

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Beijing
  - Tianjin Medical University General Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No